CLINICAL TRIAL: NCT07407166
Title: Efficacy of Immunotherapy in the First Line of Treatment of Diffuse Melanoma in Slovenia and Recognition of Prognostic and Predictive Biomarkers From Primary Tumor, Faeces and Body Fluids
Brief Title: Efficacy of First-Line Immunotherapy in Metastatic Melanoma in Slovenia and Identification of Predictive Biomarkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERID-KSOPKR-0021/2021; ERIDEK-0031/2021 (Other: Ethics Committee, Institute of Oncology Ljubljana)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Melanoma; Melanoma
Keywords: Immunotherapy; First-Line Treatment
MeSH Terms: conditions — Melanoma | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First-Line Immunotherapy (Other): Patients receiving standard-of-care first-line immunotherapy for metastatic melanoma.
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — Standard-of-care first-line immunotherapy for metastatic melanoma, including immune checkpoint inhibitors (anti-PD-1 with or without anti-CTLA-4), administered according to institutional practice.

SUMMARY:
This study evaluates the effectiveness of first-line immunotherapy in patients with metastatic melanoma treated at the Institute of Oncology Ljubljana in Slovenia. The main objectives are to assess treatment response rates, progression-free survival, and treatment safety, and to identify prognostic and predictive biomarkers associated with response to immunotherapy.

Biological samples including blood, stool, and body fluids (if available) will be collected at predefined time points and analyzed for molecular tumor markers. Imaging assessments (CT or PET/CT) will be performed before treatment initiation and during follow-up to evaluate response.

The study aims to improve identification of patient subgroups who benefit from immunotherapy and those who do not, supporting better personalized treatment strategies.

DETAILED DESCRIPTION:
Metastatic melanoma is a malignant skin cancer with significant morbidity and mortality. In recent years, immunotherapy has become a standard first-line treatment option for metastatic melanoma, but clinical benefit varies substantially among patients. Reliable prognostic and predictive biomarkers are needed to identify patients who are likely to respond to immunotherapy and those who may require alternative strategies.

This prospective study is conducted at the Institute of Oncology Ljubljana and evaluates the effectiveness of first-line immunotherapy in patients with metastatic melanoma treated in Slovenia. The primary clinical outcomes include overall response rate, progression-free survival, and safety of treatment.

Patients will undergo routine imaging examinations (CT or PET/CT of the head, chest, and abdomen) prior to the start of immunotherapy and at follow-up time points (week 4, week 12, and week 28), and additionally as clinically indicated. Imaging results will be used to evaluate disease response to treatment.

In parallel, biological samples will be collected at the same time points, including peripheral blood (10 mL), stool samples, and samples of pleural or peritoneal effusions when present. Samples will be analyzed for molecular tumor markers to explore associations with clinical response and survival outcomes.

The study aims to identify biomarker-based subgroups of patients for whom immunotherapy is beneficial and those for whom it is not, contributing to improved individualized treatment approaches in metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Metastatic (diffuse) melanoma

Planned first-line immunotherapy treatment

Signed informed consent for participation in the study

Exclusion Criteria:

Age < 18 years

Inability to provide informed consent

Any condition preventing participation or sample collection according to investigator judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) to First-Line Immunotherapy | Up to 28 weeks after start of immunotherapy
  Proportion of patients with metastatic melanoma achieving complete response (CR) or partial response (PR) during first-line immunotherapy, assessed by imaging (CT or PET/CT)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 years
  Time from initiation of first-line immunotherapy to disease progression or death from any cause.
Time to Disease Progression | Up to 3 years
  Time from initiation of first-line immunotherapy to documented disease progression assessed by imaging.
Safety of First-Line Immunotherapy | Up to 3 years
  Incidence of treatment-related adverse events during first-line immunotherapy.
Predictive and Prognostic Biomarkers in Blood, Stool and Body Fluids | Baseline and weeks 4, 12, and 28
  Identification of molecular biomarkers in blood (10 mL), stool, and pleural/peritoneal effusions (if present) associated with response to immunotherapy and survival outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia